CLINICAL TRIAL: NCT05907824
Title: Long-term Prognosis Comparison Between Parenchyma-sparing and Oncologic Resections for Non-functional Neuroendocrine Tumors of the Pancreatic Body and Tail ≤ 3cm: a Real-world Data Study
Brief Title: Long-term Prognosis for Non-functional Neuroendocrine Tumors of the Pancreatic Body and Tail ≤ 3cm
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Collaborators: The Third Affiliated Hospital of Soochow University (Other); Qilu Hospital of Shandong University (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Southern Medical University, China (Other)
Responsible Party: Principal Investigator, Xian-Jun Yu, President of Fudan University Shanghai Cancer Center, Fudan University
Other Study IDs: CSPAC-NEN-5
Record Dates: First submitted 2023-05-29; First posted 2023-06-18 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Non Functioning Pancreatic Endocrine Tumor
Keywords: Non Functioning Pancreatic Endocrine Tumor; Body and Tail of the Pancreas; Parenchyma-sparing Resection; Oncologic Resection; Long-term Prognosis
MeSH Terms: conditions — Non functioning pancreatic endocrine tumor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parenchyma-sparing Resections: Parenchyma-sparing resections, including open, laparoscopic, or robotic pancreatic enucleation, duodenum-preserving pancreatic head resection, middle segment pancreatectomy, and spleen-preserving distal pancreatectomy, without standard lymph node dissection.
  Interventions: Other: Histopathological review, long-term prognosis and quality of life follow-up
- Oncologic Resections: Oncologic resections, including open, laparoscopic, or robotic pancreaticoduodenectomy or distal pancreatectomy, with standard lymph node dissection.
  Interventions: Other: Histopathological review, long-term prognosis and quality of life follow-up

INTERVENTIONS:
Other: Histopathological review, long-term prognosis and quality of life follow-up — Histopathological review, long-term prognosis and quality of life follow-up

SUMMARY:
This study aims to quantify the malignant potential of non-functional neuroendocrine tumors of the pancreatic body and tail ≤ 3 cm by collecting real-world data from large pancreatic centers across the country, and to evaluate the appropriateness of parenchyma-sparing resection and oncologic resection.

DETAILED DESCRIPTION:
According to epidemiological investigations, the incidence of neuroendocrine tumors has increased 6.4-fold (6.98 per 100,000) . There is controversy in the latest guidelines regarding the management of sporadic non-functional pancreatic neuroendocrine tumors (pNETs) ≤ 2 cm, including follow-up and the choice between parenchyma-sparing resection (PSR) and oncologic resection (OR) . Although pNETs are generally considered indolent tumors, current experience suggests that 9.5%-12.3% of pNETs ≤ 2 cm may have lymph node metastasis, and nearly 20% of resected tumors exhibit one or more invasive features. Awareness of surgical treatment for these patients has been increasing gradually. However, there is no clear recommendation for the choice of surgical approach, and if OR is routinely performed, its prognostic value is unclear and there may be a risk of overtreatment.

The advantages of PSR include preservation of both endocrine and exocrine pancreatic function. However, the main oncological limitations of these techniques are inadequate surgical margin clearance and the risk of lack of lymph node dissection. A recent retrospective analysis of prospective databases from four large pancreatic surgery centers showed that for ≤ 3 cm non-functional pNETs, PSR or lymph node-preserving resection had less blood loss, shorter operation time, lower complications rate, and similar long-term oncological outcomes compared to OR. However, this study did not differentiate the tumor locations, as pNETs in the pancreatic head and body/tail have different lymphatic drainage patterns and surgical approaches. Furthermore, the study also showed significant differences in the proportion of PSR and the rate of positive lymph nodes between tumors located in the pancreatic head and those in the body/tail.

The ability of existing literature to provide reliable guidelines for pNETs is limited by the low incidence of the disease and short follow-up times. This study aims to quantify the malignant potential of pNETs of the pancreatic body and tail ≤ 3 cm by collecting real-world data from large pancreatic centers across the country, and to evaluate the appropriateness of PSR and OR.

ELIGIBILITY:
Inclusion Criteria:

* Non-functional neuroendocrine tumors of the pancreatic body and tail ≤ 3 cm.

Exclusion Criteria:

* Presence of liver or distant metastasis.
* Presence of concomitant malignancy.
* Multifocal or recurrent disease.
* Presence of hereditary syndrome (MEN1, VHL, NF).
* Presence of symptoms (specific symptoms of clinical syndromes suspected to be related to excessive secretion of bioactive compounds).
* History of preoperative antitumor therapy.
* Loss to follow-up.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Non-functional neuroendocrine tumors of the pancreatic body and tail ≤ 3 cm.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Through study completion, an average of 1 year.
  The time from the surgery to death from any cause.
Disease-free survival (DFS) | Through study completion, an average of 1 year.
  The time of surgery to the time of tumor recurrence or death from any cause.

SECONDARY OUTCOMES:
Perioperative complication rate | Within 90 days after surgery.
  Adverse events that occur during or after the surgery, including the incidence of postoperative complications reported according to the Clavien-Dindo classification, clinical relevant postoperative pancreatic fistula (POPF), postoperative pancreatic hemorrhage (PPH), delayed gastric emptying (DGE), reoperation rate and mortality rate within 90 days after surgery.
Postoperative pathological staging | From the date of surgery to 1 month after surgery.
  The tumor staging according to the 8th edition of the AJCC TNM staging system.
G staging | From the date of surgery to 1 month after surgery.
  The G staging evaluated according to the 2019 WHO classification and grading criteria for digestive neuroendocrine tumors.
R0 resection rate | From the date of surgery to 1 month after surgery.
  R0 margin rate on postoperative pathological assessment.
Lymph node positivity rate | From the date of surgery to 1 month after surgery.
  Lymph node positivity rate on postoperative pathological assessment.
Life quality satisfaction evaluated according to a scale. | Through study completion, an average of 1 year.
  The patient's health-related quality of life after surgical intervention. It includes physical, emotional, and social aspects of a patient's well-being. This study evaluated quality of life using a telephone survey.

CONTACTS AND LOCATIONS:
Overall Officials: Xianjun Yu, MD, PhD, Principal Investigator — Fudan University; Shunrong Ji, PhD, Study Director — Fudan University
Locations (1):
- Department of Pancreatic Surgery, Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dasari A, Shen C, Halperin D, Zhao B, Zhou S, Xu Y, Shih T, Yao JC. Trends in the Incidence, Prevalence, and Survival Outcomes in Patients With Neuroendocrine Tumors in the United States. JAMA Oncol. 2017 Oct 1;3(10):1335-1342. doi: 10.1001/jamaoncol.2017.0589. PMID 28448665
- [Background] Falconi M, Eriksson B, Kaltsas G, Bartsch DK, Capdevila J, Caplin M, Kos-Kudla B, Kwekkeboom D, Rindi G, Kloppel G, Reed N, Kianmanesh R, Jensen RT; Vienna Consensus Conference participants. ENETS Consensus Guidelines Update for the Management of Patients with Functional Pancreatic Neuroendocrine Tumors and Non-Functional Pancreatic Neuroendocrine Tumors. Neuroendocrinology. 2016;103(2):153-71. doi: 10.1159/000443171. Epub 2016 Jan 5. No abstract available. PMID 26742109
- [Background] Halfdanarson TR, Strosberg JR, Tang L, Bellizzi AM, Bergsland EK, O'Dorisio TM, Halperin DM, Fishbein L, Eads J, Hope TA, Singh S, Salem R, Metz DC, Naraev BG, Reidy-Lagunes DL, Howe JR, Pommier RF, Menda Y, Chan JA. The North American Neuroendocrine Tumor Society Consensus Guidelines for Surveillance and Medical Management of Pancreatic Neuroendocrine Tumors. Pancreas. 2020 Aug;49(7):863-881. doi: 10.1097/MPA.0000000000001597. PMID 32675783
- [Background] Gratian L, Pura J, Dinan M, Roman S, Reed S, Sosa JA. Impact of extent of surgery on survival in patients with small nonfunctional pancreatic neuroendocrine tumors in the United States. Ann Surg Oncol. 2014 Oct;21(11):3515-21. doi: 10.1245/s10434-014-3769-4. Epub 2014 May 20. PMID 24841347
- [Background] Xu JZ, Wang WQ, Zhang SR, Xu HX, Wu CT, Qi ZH, Gao HL, Ni QX, Liu L, Yu XJ. Intrinsic Contact Between T and N Classifications in Resected Well-Moderately Differentiated Locoregional Pancreatic Neuroendocrine Neoplasms. Ann Surg Oncol. 2018 Mar;25(3):647-654. doi: 10.1245/s10434-017-6289-1. Epub 2017 Dec 12. PMID 29235006
- [Background] Tanaka M, Heckler M, Mihaljevic AL, Probst P, Klaiber U, Heger U, Schimmack S, Buchler MW, Hackert T. Systematic Review and Metaanalysis of Lymph Node Metastases of Resected Pancreatic Neuroendocrine Tumors. Ann Surg Oncol. 2021 Mar;28(3):1614-1624. doi: 10.1245/s10434-020-08850-7. Epub 2020 Jul 27. PMID 32720049
- [Background] Partelli S, Massironi S, Zerbi A, Niccoli P, Kwon W, Landoni L, Panzuto F, Tomazic A, Bongiovanni A, Kaltsas G, Sauvanet A, Bertani E, Mazzaferro V, Caplin M, Armstrong T, Weickert MO, Ramage J, Segelov E, Butturini G, Staettner S, Cives M, Frilling A, Moulton CA, He J, Boesch F, Selberheer A, Twito O, Castaldi A, De Angelis CG, Gaujoux S, Holzer K, Wilson CH, Almeamar H, Vigia E, Muffatti F, Luca M, Lania A, Ewald J, Kim H, Salvia R, Rinzivillo M, Smid A, Gardini A, Tsoli M, Hentic O, Colombo S, Citterio D, Toumpanakis C, Ramsey E, Randeva HS, Srirajaskanthan R, Croagh D, Regi P, Gasteiger S, Invernizzi P, Ridolfi C, Giovannini M, Jang JY, Bassi C, Falconi M. Management of asymptomatic sporadic non-functioning pancreatic neuroendocrine neoplasms no larger than 2 cm: interim analysis of prospective ASPEN trial. Br J Surg. 2022 Nov 22;109(12):1186-1190. doi: 10.1093/bjs/znac267. No abstract available. PMID 35986682
- [Background] Partelli S, Mazza M, Andreasi V, Muffatti F, Crippa S, Tamburrino D, Falconi M. Management of small asymptomatic nonfunctioning pancreatic neuroendocrine tumors: Limitations to apply guidelines into real life. Surgery. 2019 Aug;166(2):157-163. doi: 10.1016/j.surg.2019.04.003. Epub 2019 May 17. PMID 31109657
- [Background] Chivukula SV, Tierney JF, Hertl M, Poirier J, Keutgen XM. Operative resection in early stage pancreatic neuroendocrine tumors in the United States: Are we over- or undertreating patients? Surgery. 2020 Jan;167(1):180-186. doi: 10.1016/j.surg.2019.04.061. Epub 2019 Sep 16. PMID 31537303
- [Background] Pea A, Tanno L, Nykanen T, Prasad P, Tuncer C, Robinson S, Marchegiani G. Comparison of Oncological and Surgical Outcomes Between Formal Pancreatic Resections and Parenchyma-Sparing Resections for Small PanNETs (<2 cm): Pancreas2000 Research and Educational Program (Course 9) Study Protocol. Front Med (Lausanne). 2020 Sep 10;7:559. doi: 10.3389/fmed.2020.00559. eCollection 2020. PMID 33015105
- [Background] Nesti C, Brautigam K, Benavent M, Bernal L, Boharoon H, Botling J, Bouroumeau A, Brcic I, Brunner M, Cadiot G, Camara M, Christ E, Clerici T, Clift AK, Clouston H, Cobianchi L, Cwikla JB, Daskalakis K, Frilling A, Garcia-Carbonero R, Grozinsky-Glasberg S, Hernando J, Hervieu V, Hofland J, Holmager P, Inzani F, Jann H, Jimenez-Fonseca P, Kacmaz E, Kaemmerer D, Kaltsas G, Klimacek B, Knigge U, Kolasinska-Cwikla A, Kolb W, Kos-Kudla B, Kunze CA, Landolfi S, La Rosa S, Lopez CL, Lorenz K, Matter M, Mazal P, Mestre-Alagarda C, Del Burgo PM, van Dijkum EJMN, Oleinikov K, Orci LA, Panzuto F, Pavel M, Perrier M, Reims HM, Rindi G, Rinke A, Rinzivillo M, Sagaert X, Satiroglu I, Selberherr A, Siebenhuner AR, Tesselaar MET, Thalhammer MJ, Thiis-Evensen E, Toumpanakis C, Vandamme T, van den Berg JG, Vanoli A, van Velthuysen MF, Verslype C, Vorburger SA, Lugli A, Ramage J, Zwahlen M, Perren A, Kaderli RM. Hemicolectomy versus appendectomy for patients with appendiceal neuroendocrine tumours 1-2 cm in size: a retrospective, Europe-wide, pooled cohort study. Lancet Oncol. 2023 Feb;24(2):187-194. doi: 10.1016/S1470-2045(22)00750-1. Epub 2023 Jan 11. PMID 36640790
- [Background] Bolm L, Nebbia M, Wei AC, Zureikat AH, Fernandez-Del Castillo C, Zheng J, Pulvirenti A, Javed AA, Sekigami Y, Petruch N, Qadan M, Lillemoe KD, He J, Ferrone CR; PAncreatic Neuroendocrine Disease Alliance (PANDA). Long-term Outcomes of Parenchyma-sparing and Oncologic Resections in Patients With Nonfunctional Pancreatic Neuroendocrine Tumors <3 cm in a Large Multicenter Cohort. Ann Surg. 2022 Sep 1;276(3):522-531. doi: 10.1097/SLA.0000000000005559. Epub 2022 Jun 27. PMID 35758433
- [Background] Tsuchikawa T, Tanaka K, Nakanishi Y, Asano T, Noji T, Nakamura T, Okamura K, Shichinohe T, Hirano S. Clinical Impact of Organ-Preserving Surgery for Pancreatic Neuroendocrine Neoplasms: A Single-Center Experience. Pancreas. 2021 Feb 1;50(2):196-200. doi: 10.1097/MPA.0000000000001739. PMID 33565795